CLINICAL TRIAL: NCT02256384
Title: Evaluation of Respiratory Acoustic Monitor in Children After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Masimo Corporation (Industry); Children's Medical Center Dallas (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-6421
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Complications; Pediatric
Keywords: Respiration Rate; Respiratory Acoustic Monitor; postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory Acoustic Monitoring (Experimental): All participants will wear the respiratory acoustic monitoring device.
  Interventions: Device: Respiratory Acoustic Monitor

INTERVENTIONS:
Device: Respiratory Acoustic Monitor — Examine the reliability and accuracy of the respiratory acoustic monitor.

SUMMARY:
The study will evaluate the performance of measuring respiration rate with the Respiratory Acoustic Monitoring (RAM).

DETAILED DESCRIPTION:
The study seeks to determine the reliability and accuracy of the acoustic respiratory monitoring (RAM) in comparison of clinically completed transthoracic impedance monitoring (TI) and manual counting of respiratory rate in postoperative pediatric patients at risk of adverse respiratory events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children 2 to 16 years of age
* In-patients or 23 hour short stay patients who had a tonsillectomy with a diagnosis or symptoms of obstructive sleep apnea or who had any surgery and receiving an opioid by patient controlled analgesia for post-operative pain control
* Child weighs at least 10 kg on day of surgery

Exclusion Criteria:

* Patient has skin abnormalities (rash, eczema, etc.) at the planned application sites that would interfere with sensor or electrode applications.
* Patient is admitted to the Intensive Care Unit
* Patient has tracheostomy
* Patient is on non-invasive ventilator support

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Patino, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Peter Szmuk, MD, Principal Investigator — UT Southwestern Medical Center- Dallas
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UT Southwestern Medical Center - Dallas, Dallas, Texas

REFERENCES:
- [Result] Patino M, Kalin M, Griffin A, Minhajuddin A, Ding L, Williams T, Ishman S, Mahmoud M, Kurth CD, Szmuk P. Comparison of Postoperative Respiratory Monitoring by Acoustic and Transthoracic Impedance Technologies in Pediatric Patients at Risk of Respiratory Depression. Anesth Analg. 2017 Jun;124(6):1937-1942. doi: 10.1213/ANE.0000000000002062. PMID 28448390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Whenever possible, the family will be approached at a pre-surgical clinic visit or contacted by phone the day before recruitment to explain the study. Consent will occur in person at either a clinic visit prior to the day of surgery, in the pre-operative area on the day of surgery, or in the patient's room after surgery.
Groups:
- Respiratory Acoustic Monitoring: All participants will wear the respiratory acoustic monitoring device. Respiratory Acoustic Monitor: Examine the reliability and accuracy of the respiratory acoustic monitor.
Period: Overall Study
Arm/Group | Respiratory Acoustic Monitoring
Started | 76
Completed | 62
Not Completed | 14
Not completed — Withdrawal by Subject | 12
Not completed — Equipment not capturing data | 2

BASELINE CHARACTERISTICS:
Arm/Group | Respiratory Acoustic Monitoring
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Reliability/ Accuracy of Respiratory Acoustic Monitoring (RAM)
Description: The respiratory acoustic monitor records three vital signs: Respiration rate recorded in breaths per minute, oxygen saturation recorded in percentage, and heart rate recorded in beats per minute.
  The reliability and accuracy of the respiratory data collected by the RAM was examined by comparing to data collected clinically by the manual counting of the respiratory rate and by the respiratory rate measure by transthoracic impedance . The accuracy of RAM was examined when a staff member goes and register these measurements that occur simultaneously during the first minute of every 2 hour interval to a maximum of a 24 hour monitoring time.
Time Frame: Up to 24 hours after surgery
Population: 62 children from 2 to 16 years old that required postoperatory admission for continuous respiratory monitoring.The respiratory rate was measured and recorded at the same time every 2 hours from the: (a) RAM monitor, (b) thoracic impedance, and (c) manual count over 1 minute. In addition the presence of alarms was also recorded.
Measure: Mean (Standard Error); unit: Breaths per minute
Groups:
- Manual Counting: Respiratory rate was recorded by clinical evaluation every 2 hours during the first minute of the evaluation and recorded also simultaneously by RAM and by transthoracic impedance.
- Transthoracic Impedance: The respiratory rate was measured by Transthoracic impedance with the use of the electrocardiogram pads.
Arm/Group | Respiratory Acoustic Monitoring | Manual Counting | Transthoracic Impedance
Number analyzed (Participants) | 62 | 62 | 62
Breaths per minute | 19.7 (0.52) | 19.6 (0.56) | 21.3 (0.77)

2. Secondary Outcome: Presence of False Alarms
Description: To evaluate the presence of false alarms, bedside clinical monitoring was done every two hour during 5 to 15 minutes (random sample) recording the respiratory rates and evaluating the presence of alarms. If an alarm was activated during the bedside monitoring, it was verified by the investigator if the respiratory rate provided by the device was consistent with the clinical evaluation. False alarms were considered those alarms that are triggered by the device, but during simultaneous clinical evaluation it was verified that the number of breaths per minute were inaccurate. Therefore, the higher number of false alarms detected by one type of monitoring indicates that the device is less reliable detecting the respiratory rate.
Time Frame: Up to 24 hours after surgery
Population: The presence of alarms and their evaluation as true or false was recorded during 5 to 15 minutes of a fixed interval of every 2 hours.
Measure: Mean (Standard Deviation); unit: Number of false alarms per patient
Groups:
- Respiratory Acoustic Monitoring: All participants wore the respiratory acoustic monitoring device. Respiratory Acoustic Monitor: Examine the reliability and accuracy of the respiratory acoustic monitor.
- Transthoracic Impedance: All participants wore continuous electrocardiographic monitoring capable of recording respiratory rate continuously and the alarm was set up by defaulted respiratory alarms already selected during the regular clinical practice.
Arm/Group | Respiratory Acoustic Monitoring | Transthoracic Impedance
Number analyzed (Participants) | 62 | 62
Number of false alarms per patient | 0.18 (0.71) | 1.00 (2.78)

3. Secondary Outcome: Tolerance of the RAM
Description: The tolerance is defined as the ratio of the time the sensor stays in place divided by the total expected time of monitoring, expressed as a percentage. The tolerance to the transthoracic impedance pads was not evaluated during this study considering that this is the standard monitoring and that is usually tolerated during the total expected time of monitoring.
Time Frame: Up to 24 hours after surgery
Measure: Mean (Standard Error); unit: percentage of time sensor stays in place
Arm/Group | Respiratory Acoustic Monitoring
Number analyzed (Participants) | 62
percentage of time sensor stays in place | 87 (4.26)

ADVERSE EVENTS:
Description: No serious adverse events were reported related to wearing the monitor sensors. Information regarding skin irritation due to the placement of the sensor was collected just by one of the institutions involved in the study, but was not recorded by the other institution. The total number of participants recruited at the institution that reports the incidence of skin irritation were 30 participants.
Arm/Group | Respiratory Acoustic Monitoring
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Respiratory Acoustic Monitoring (N=30)
Skin irritation (Skin and subcutaneous tissue disorders) | 4 — Participants complained of their skin being irritated by the adhesive that is used on the sensors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No